CLINICAL TRIAL: NCT00846729
Title: Preserving Renal Longevity in Living Kidney Donors
Brief Title: Comparative Renal Function of Young (18-45 Years) and Ageing (55 Years and Above) Kidney Donors
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jane C. Tan, Associate Professor of Medicine (Nephrology), Stanford University
Other Study IDs: SU-02092009-1778; IRB eProtocol #13584; SPO 45339
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood samples are obtained throughout the kidney function study. These samples are analyzed for Iothalamate and PAH (markers of kidney function) only.
  2. Kidney tissue obtained by biopsy at the time of surgery are used to analyze the structure of the kidney.
  No Tissue or Blood is used for genetic analysis.

INTERVENTIONS:
Procedure: CT angiogram of the remaining kidney.
Procedure: Kidney Function study using Iothalamate & PAH as clearance markers

SUMMARY:
It is our purpose in this study to compare the kidney structure and function of older patients to that of young patients before and after removal of a single kidney for transplant donation and to examine the remaining kidney's ability to adapt and maintain function over time. More specifically, we aim to examine the effect of uninephrectomy on adaptive hyperfiltration in the remaining kidney. A secondary aim is to investigate whether subjects in the aging population undergo compensation to the same extent as younger subjects. We will also examine the compensatory rise in GFR (glomerular filtration rate) that follows uninephrectomy in both groups, and, again, compare the results in the aged versus young subjects. This will help in delineating the extent to which the aging population can be a potential source of living kidney donors for kidney transplantation.

It is also our purpose with this study to refine the tests to be used in the donor evaluation process so as to accurately identify ideal candidates for safe kidney donation.

DETAILED DESCRIPTION:
Screening Procedures: Patients will be identified after acceptance by Stanford's kidney transplant team as appropriate candidates for living kidney donation prior to their surgery.

The following assessments will be performed over the course of 4 years for this protocol.

A. Informed Consent will be obtained.

B. A Cimetidine Blocked 24 hour urine collection will be obtained prior to surgery.

C. DETAILED KIDNEY FUNCTION STUDIES will be performed using iothalamate, and PAH at three different times:

1. Prior to surgery for uninephrectomy (the night before to months before surgery)
2. 6 months to 1 year post kidney donation.
3. 4 years after kidney donation.

D. The Structure of the Kidney will also be assessed at three different times during this protocol:

1. Cortical and whole kidney volumes will be determined using the clinical MRI or CT performed routinely for kidney donor evaluation.
2. At the time of surgery, in the operating room: A single wedge biopsy of the kidney will be taken for morphometric and later genetic analysis. *NOTE: Genetic analysis is for the genetics of ageing not disease. In this procedure, a small wedge kidney biopsy is excised under direct visualization by the transplant surgeon after the kidney has been removed from the donor and before the kidney is transplanted into the recipient. The area of excision is then oversewn and checked for bleeding.

   The size (volume) of the Tx kidney will be measured by water displacement in a graduated cylinder immediately before Tx. This volume will be used in our calculations to estimate the number of glomeruli in youthful vs ageing kidneys.
3. A second MRI or CT will be obtained 6 months to 1 year after kidney donation to measure the kidney's overall compensatory growth and increase in cortical volume for comparison with the pre-operative volumes.

ELIGIBILITY:
Inclusion Criteria:1. Patients who are over the age of 18. 2. Patients who are undergoing surgical uninephrectomy for the purpose of living donation for transplantation 3. Adults who had a single kidney removed for transplant donation 10-20 years ago.

4. All Patients enrolled in this study must be between the ages of 18 and 45 years or 55 years or older.

5. Patients undergoing surgery for kidney donation who exhibit mild hypertension controlled with one medication. Any age accepted Exclusion Criteria:1. Patients under the age of 18.

2. Patients between the ages of 46 and 54 3. Patients who are allergic to Inulin, Iothalamate, or PAH. 4. Women who are pregnant. 5. Other "Vulnerable Subjects"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Men and Women who are undergoing surgery for kidney donation for transplantation who are between the ages of 18 and 45, and 55 and above.
  2. Men and women who are undergoing surgery for kidney donation for transplantation who exhibit mild hypertension.
  3. Men and women who donated a kidney for transplantation 10 to 20 years ago.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2003-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Diminished adaptive response to living kidney donation in ageing donors as compared to living donors. | 4 years

SECONDARY OUTCOMES:
Renal Failure & new onset, or worsening, of hypertension in living kidney donors | 4 yr

CONTACTS AND LOCATIONS:
Overall Officials: Bryan D Myers, Principal Investigator — Stanford University; Jane C. Tan, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States